CLINICAL TRIAL: NCT01571596
Title: An Open-Label, Long-Term, Extension Study to Evaluate the Safety and Efficacy of KRN23 in Adult Subjects With X-Linked Hypophosphatemia
Brief Title: An Extension Study of KRN23 in Adults With X-Linked Hypophosphatemia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Kyowa Kirin Co., Ltd. (Industry)
Collaborators: Kyowa Hakko Kirin Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KRN23-INT-002
Record Dates: First submitted 2012-02-23; First posted 2012-04-05 (Estimated); Results first posted 2021-02-17 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: X-linked Hypophosphatemia
Keywords: XLH
MeSH Terms: conditions — Familial Hypophosphatemic Rickets | interventions — burosumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- KRN23 (Experimental): Escalating doses of KRN23 (0.05, 0.10, 0.30, and 0.60 mg/kg) will be administered SC every 28 days (up to 12 doses)
  Interventions: Drug: KRN23

INTERVENTIONS:
Drug: KRN23 — Subjects will receive escalating doses of KRN23 administered by SC injection every 28-days (up to 12 doses) based on a dosing algorithm and discretion of Investigator and Sponsor.

SUMMARY:
The primary purpose of this study is to assess the safety and efficacy of repeated subcutaneous (SC) injections of KRN23 in adult subjects with X-Linked Hypophosphatemia (XLH).

ELIGIBILITY:
Inclusion Criteria:

1. Satisfactory completion of KKP's sponsored KRN23-INT-001 clinical trial
2. eGFR ≥ 60 mL/min
3. Corrected Ca < 10.8 mg/dL
4. For female of child-bearing potential, a negative serum pregnancy test
5. A willingness to utilize adequate contraception and not become pregnant [or to have their partner(s) become pregnant] during the study
6. Additional inclusion criteria apply

Exclusion Criteria:

1. Subject experienced a safety-related event in the KRN23-INT-001 study
2. Pregnant or lactating female subject or pregnant or female planning to become pregnant during the study
3. Receipt of a live (attenuated) vaccine (except for influenza vaccines) during the course of the KRN23-INT-001 study and/or of this study
4. Condition which could present a concern for either the subject's safety or difficulty with data interpretation
5. Additional exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2012-02; Primary Completion 2013-09 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amy Zhang, PhD, Study Director — Kyowa Hakko Kirin Pharma, Inc.
Locations (6):
- United States (5):
  - University of California San Francisco, San Francisco, California
  - Yale University School of Medicine, New Haven, Connecticut
  - Clinical Research Center, Indiana University School of Medicine, Indianapolis, Indiana
  - Duke Clinical Research Unit, Durham, North Carolina
  - University of Texas Health Science Center at Houston, Houston, Texas
- Shriners Hospital for Children - Canada, Montreal, Quebec, Canada

REFERENCES:
- [Derived] Imel EA, Zhang X, Ruppe MD, Weber TJ, Klausner MA, Ito T, Vergeire M, Humphrey JS, Glorieux FH, Portale AA, Insogna K, Peacock M, Carpenter TO. Prolonged Correction of Serum Phosphorus in Adults With X-Linked Hypophosphatemia Using Monthly Doses of KRN23. J Clin Endocrinol Metab. 2015 Jul;100(7):2565-73. doi: 10.1210/jc.2015-1551. Epub 2015 Apr 28. PMID 25919461
- See also: Related Info — http://www.clinicaltrials.gov/ct2/show/NCT00830674?term=XLH&rank=1
- See also: Related Info — http://www.clinicaltrials.gov/ct2/show/NCT01340482?term=KRN23&rank=1

RESULTS

PARTICIPANT FLOW:
Groups:
- Bone Substudy KRN23; Bone Substudy Placebo: A Bone substudy in eligible subjects will evaluate the effects of KRN23 on various bone parameters. Subjects will undergo clinical assessments, inclusive of DXA and pQCT at Visits 17 and 33 (prior to dosing), and the end-of-study visit, Visit 49. A subset of subjects will have a bone biopsy of the iliac crest at Visit 33.
Period: Overall Study
Arm/Group | KRN23 | Bone Substudy KRN23 | Bone Substudy Placebo
Started | 21 | 1 | 1
Completed | 19 | 0 | 0
Not Completed | 2 | 1 | 1
Not completed — Adverse Event | 2 | 0 | 0
Not completed — Study Terminated by the Sponsor | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | KRN23 | Bone Substudy KRN23 | Bone Substudy Placebo | Total
Number analyzed (Participants) | 21 | 1 | 1 | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 20 | 1 | 1 | 22
  >=65 years | 1 | 0 | 0 | 1
Age, Continuous [Mean (Full Range); unit: years] | 43.0 [19 to 66] | 22 [22 to 22] | 28 [28 to 28] | 41.1 [19 to 66]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 1 | 1 | 14
  Male | 9 | 0 | 0 | 9
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White/Caucasian | 20 | 1 | 1 | 22
  Black/African American/African Caribbean | 1 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  Canada | 0 | 1 | 1 | 2
  United States | 21 | 0 | 0 | 21

OUTCOME MEASURES:

1. Primary Outcome: Safety and Efficacy of Repeated SC Injections of KRN23.
Description: Safety and efficacy of repeated SC injections of KRN23, from Baseline, as assessed by serum phosphorus levels, immunogenicity, adverse events and clinically significant changes in vital signs and laboratory testing.
Time Frame: 13.5 months,(50 visits)
Measure: Count of Participants; unit: Participants
Arm/Group | KRN23 | Bone Substudy KRN23 | Bone Substudy Placebo
Number analyzed (Participants) | 21 | 1 | 1
Participants
  With Any TEAE | 21 | 1 | 1
  With Any Drug-related TEAE | 13 | 1 | 0
  With Any TEAE with an Outcome of Death | 0 | 0 | 0
  With Any Serious TEAE | 3 | 0 | 0
  With Any Drug-related Serious TEAE | 0 | 0 | 0
  With Any Serious TEAE with an Outcome of Death | 0 | 0 | 0

2. Secondary Outcome: Evaluation of Effect of Repeated SC Injections of KRN23
Description: Effect of repeated SC injections of KRN23, from baseline, on pharmacodynamic parameters (serum phosphorus)
Time Frame: 13.5 months, (50 visits)
Population: Efficacy analysis set: All subjects who received at least 1 dose of KRN23 and completed at least one 28-day post-dose evaluation.
Measure: Mean (Full Range); unit: mg/dL
Arm/Group | KRN23
Number analyzed (Participants) | 22
mg/dL
  Baseline | 1.85 [1.2 to 2.3]
  Ext Visit 1 /0: number analyzed (Participants) | 21
  Ext Visit 1 /0 | 1.88 [1.3 to 2.5]
  Ext Visit 2 /7 | 2.86 [2.1 to 3.6]
  Ext Visit 3 /14 | 2.87 [2.0 to 3.5]
  Ext Visit 4 /25 | 2.48 [2.0 to 3.0]
  Ext Visit 5 /0: number analyzed (Participants) | 21
  Ext Visit 5 /0 | 2.25 [1.8 to 3.1]
  Ext Visit 6 /7: number analyzed (Participants) | 21
  Ext Visit 6 /7 | 2.91 [2.1 to 3.9]
  Ext Visit 7 /14: number analyzed (Participants) | 21
  Ext Visit 7 /14 | 2.95 [2.3 to 3.8]
  Ext Visit 8 /25: number analyzed (Participants) | 20
  Ext Visit 8 /25 | 2.67 [1.9 to 3.3]
  Ext Visit 9 /0: number analyzed (Participants) | 21
  Ext Visit 9 /0 | 2.43 [1.6 to 2.9]
  Ext Visit 10 /7: number analyzed (Participants) | 21
  Ext Visit 10 /7 | 2.96 [2.2 to 3.8]
  Ext Visit 11 /14: number analyzed (Participants) | 21
  Ext Visit 11 /14 | 2.84 [2.2 to 3.5]
  Ext Visit 12 /25: number analyzed (Participants) | 21
  Ext Visit 12 /25 | 2.59 [2.1 to 3.5]
  Ext Visit 13 /0: number analyzed (Participants) | 21
  Ext Visit 13 /0 | 2.42 [1.7 to 3.1]
  Ext Visit 14 /7: number analyzed (Participants) | 21
  Ext Visit 14 /7 | 2.92 [1.9 to 3.8]
  Ext Visit 15 /14: number analyzed (Participants) | 21
  Ext Visit 15 /14 | 2.90 [2.1 to 3.6]
  Ext Visit 16 /25: number analyzed (Participants) | 21
  Ext Visit 16 /25 | 2.57 [1.9 to 3.4]
  Ext Visit 17 /0: number analyzed (Participants) | 20
  Ext Visit 17 /0 | 2.35 [1.7 to 3.4]
  Ext Visit 18 /7: number analyzed (Participants) | 20
  Ext Visit 18 /7 | 2.82 [2.1 to 3.5]
  Ext Visit 19 /14: number analyzed (Participants) | 21
  Ext Visit 19 /14 | 2.74 [2.0 to 3.5]
  Ext Visit 20 /25: number analyzed (Participants) | 21
  Ext Visit 20 /25 | 2.60 [1.8 to 3.5]
  Ext Visit 21 /0: number analyzed (Participants) | 20
  Ext Visit 21 /0 | 2.35 [1.7 to 3.0]
  Ext Visit 22 /7: number analyzed (Participants) | 20
  Ext Visit 22 /7 | 2.94 [2.3 to 3.8]
  Ext Visit 23 /14: number analyzed (Participants) | 19
  Ext Visit 23 /14 | 2.93 [2.0 to 3.8]
  Ext Visit 24 /25: number analyzed (Participants) | 20
  Ext Visit 24 /25 | 2.60 [1.8 to 3.5]
  Ext Visit 25 /0: number analyzed (Participants) | 20
  Ext Visit 25 /0 | 2.37 [1.8 to 2.9]
  Ext Visit 26 /7: number analyzed (Participants) | 20
  Ext Visit 26 /7 | 2.83 [2.3 to 3.5]
  Ext Visit 27 /14: number analyzed (Participants) | 19
  Ext Visit 27 /14 | 2.79 [2.1 to 3.5]
  Ext Visit 28 /25: number analyzed (Participants) | 20
  Ext Visit 28 /25 | 2.59 [2.1 to 3.2]
  Ext Visit 29 /0: number analyzed (Participants) | 20
  Ext Visit 29 /0 | 2.41 [1.7 to 3.4]
  Ext Visit 30 /7: number analyzed (Participants) | 18
  Ext Visit 30 /7 | 2.87 [2.1 to 3.7]
  Ext Visit 31 /14: number analyzed (Participants) | 18
  Ext Visit 31 /14 | 2.81 [1.9 to 3.5]
  Ext Visit 32 /25: number analyzed (Participants) | 19
  Ext Visit 32 /25 | 2.55 [2.0 to 3.4]
  Ext Visit 33 /0: number analyzed (Participants) | 18
  Ext Visit 33 /0 | 2.42 [1.6 to 3.2]
  Ext Visit 34 /7: number analyzed (Participants) | 18
  Ext Visit 34 /7 | 2.79 [2.0 to 3.8]
  Ext Visit 35 /14: number analyzed (Participants) | 17
  Ext Visit 35 /14 | 2.75 [1.7 to 3.4]
  Ext Visit 36 /25: number analyzed (Participants) | 19
  Ext Visit 36 /25 | 2.53 [1.9 to 3.6]
  Ext Visit 37 /0: number analyzed (Participants) | 19
  Ext Visit 37 /0 | 2.52 [1.9 to 3.4]
  Ext Visit 38 /7: number analyzed (Participants) | 19
  Ext Visit 38 /7 | 2.85 [1.9 to 3.9]
  Ext Visit 39 /14: number analyzed (Participants) | 19
  Ext Visit 39 /14 | 2.69 [1.7 to 3.7]
  Ext Visit 40 /25: number analyzed (Participants) | 19
  Ext Visit 40 /25 | 2.48 [1.8 to 3.5]
  Ext Visit 41 /0: number analyzed (Participants) | 19
  Ext Visit 41 /0 | 2.29 [1.8 to 3.2]
  Ext Visit 42 /7: number analyzed (Participants) | 19
  Ext Visit 42 /7 | 2.71 [1.7 to 3.8]
  Ext Visit 43 /14: number analyzed (Participants) | 19
  Ext Visit 43 /14 | 2.70 [2.0 to 3.6]
  Ext Visit 44 /25: number analyzed (Participants) | 19
  Ext Visit 44 /25 | 2.43 [1.9 to 2.9]
  Ext Visit 45 /0: number analyzed (Participants) | 19
  Ext Visit 45 /0 | 2.25 [1.7 to 2.8]
  Ext Visit 46 /7: number analyzed (Participants) | 19
  Ext Visit 46 /7 | 2.73 [2.1 to 3.6]
  Ext Visit 47 /14: number analyzed (Participants) | 19
  Ext Visit 47 /14 | 2.61 [1.9 to 3.4]
  Ext Visit 48 /25: number analyzed (Participants) | 19
  Ext Visit 48 /25 | 2.43 [1.9 to 3.0]
  Ext Visit 49 /38: number analyzed (Participants) | 19
  Ext Visit 49 /38 | 2.07 [1.6 to 2.6]
  Ext Visit 50 /81: number analyzed (Participants) | 4
  Ext Visit 50 /81 | 1.78 [1.6 to 1.9]

3. Other Pre Specified Outcome: Evaluation of Effect of Repeated SC Injections of KRN23 in Bone Substudy
Description: Evaluation of effect of repeated SC injections of KRN23, compared to Placebo on bone mineral density, bone quality and histomorphometric parameters.
Time Frame: 13.5 months,(50 visits)
Measure: Number; unit: units on a scale
Arm/Group | Bone Substudy KRN23 | Bone Substudy Placebo
Number analyzed (Participants) | 1 | 1
units on a scale | NA — insufficient number of participants | NA — insufficient number of participants

ADVERSE EVENTS:
Time Frame: After the first dose of study drug in study through the end of study, up to 13.5 months
Arm/Group | KRN23 | Bone Substudy KRN23 | Bone Substudy Placebo
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/1 | 0/1
Serious Adverse Events (participants affected / at risk) | 3/21 | 0/1 | 0/1
Other Adverse Events (participants affected / at risk) | 21/21 | 1/1 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | KRN23 (N=21) | Bone Substudy KRN23 (N=1) | Bone Substudy Placebo (N=1)
Cervical Spinal Stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Hypertensive crisis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | KRN23 (N=21) | Bone Substudy KRN23 (N=1) | Bone Substudy Placebo (N=1)
BRADYCARDIA (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
PALPITATIONS (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
EAR PAIN (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
VERTIGO (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
DEAFNESS (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
HYPOACUSIS (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
DRY EYE (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
EYE PRURITUS (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
VOMITING (Gastrointestinal disorders) | 1 (3) | 0 (0) | 0 (0)
GINGIVAL ULCERATION (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
TOOTHACHE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0)
LIP ULCERATION (Gastrointestinal disorders) | 0 (0) | 1 (4) | 0 (0)
NAUSEA (Gastrointestinal disorders) | 2 (4) | 0 (0) | 0 (0)
POOR DENTAL CONDITION (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
ABDOMINAL PAIN (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
LIP BLISTER (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
FOOD POISONING (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
ABDOMINAL DISCOMFORT (Gastrointestinal disorders) | 4 (6) | 0 (0) | 0 (0)
DIARRHOEA (Gastrointestinal disorders) | 3 (5) | 0 (0) | 0 (0)
IRRITABLE BOWEL SYNDROME (Gastrointestinal disorders) | 1 (10) | 0 (0) | 0 (0)
HAEMATOCHEZIA (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
INJECTION SITE HAEMATOMA (General disorders) | 0 (0) | 1 (1) | 0 (0)
INFLUENZA LIKE ILLNESS (General disorders) | 1 (1) | 0 (0) | 0 (0)
INJECTION SITE ERYTHEMA (General disorders) | 1 (1) | 0 (0) | 0 (0)
FATIGUE (General disorders) | 3 (3) | 0 (0) | 0 (0)
INJECTION SITE PAIN (General disorders) | 1 (1) | 1 (6) | 0 (0)
GRAVITATIONAL OEDEMA (General disorders) | 1 (1) | 0 (0) | 0 (0)
HYPOTHERMIA (General disorders) | 1 (1) | 0 (0) | 0 (0)
APPLICATION SITE REACTION (General disorders) | 1 (1) | 0 (0) | 0 (0)
PAIN (General disorders) | 1 (2) | 0 (0) | 0 (0)
NODULE (General disorders) | 1 (1) | 0 (0) | 0 (0)
INJECTION SITE REACTION (General disorders) | 5 (26) | 0 (0) | 0 (0)
INJECTION SITE RASH (General disorders) | 1 (1) | 0 (0) | 0 (0)
INJECTION SITE PRURITUS (General disorders) | 1 (2) | 0 (0) | 0 (0)
HEPATIC STEATOSIS (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
SEASONAL ALLERGY (Immune system disorders) | 2 (2) | 0 (0) | 0 (0)
VULVOVAGINAL MYCOTIC INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
VIRAL PHARYNGITIS (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
VIRAL INFECTION (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
URINARY TRACT INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
TOOTH INFECTION (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
SINUSITIS (Infections and infestations) | 6 (7) | 0 (0) | 0 (0)
RESPIRATORY TRACT INFECTION VIRAL (Infections and infestations) | 2 (3) | 0 (0) | 0 (0)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
POST PROCEDURAL INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
TOOTH ABSCESS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
VAGINITIS BACTERIAL (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
PHARYNGITIS STREPTOCOCCAL (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
PHARYNGITIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
NASOPHARYNGITIS (Infections and infestations) | 2 (3) | 1 (1) | 1 (1)
LARYNGITIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
INFLUENZA (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
EAR INFECTION (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
GASTROENTERITIS VIRAL (Infections and infestations) | 3 (3) | 0 (0) | 0 (0)
BRONCHITIS (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
GASTROENTERITIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
MUSCLE STRAIN (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
HEAD INJURY (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
GINGIVAL INJURY (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
EXCORIATION (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
CONTUSION (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 0 (0)
TOOTH FRACTURE (Injury, poisoning and procedural complications) | 3 (3) | 0 (0) | 0 (0)
SOFT TISSUE INJURY (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
PROCEDURAL PAIN (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
POST PROCEDURAL SWELLING (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
WHITE BLOOD CELL COUNT DECREASED (Investigations) | 1 (1) | 0 (0) | 0 (0)
NEUTROPHIL COUNT DECREASED (Investigations) | 1 (1) | 0 (0) | 0 (0)
BLOOD PRESSURE DECREASED (Investigations) | 1 (1) | 0 (0) | 0 (0)
BLOOD CREATINE PHOSPHOKINASE INCREASED (Investigations) | 1 (1) | 0 (0) | 0 (0)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 1 (2) | 0 (0) | 0 (0)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 1 (2) | 0 (0) | 0 (0)
TENDONITIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0) | 0 (0)
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0)
MUSCULOSKELETAL DISCOMFORT (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 2 (6) | 0 (0) | 0 (0)
JOINT SWELLING (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0)
JOINT EFFUSION (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
JOINT CREPITATION (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0)
HAEMARTHROSIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
CERVICAL SPINAL STENOSIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 5 (6) | 0 (0) | 0 (0)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 6 (10) | 0 (0) | 0 (0)
SYNCOPE (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
SINUS HEADACHE (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
SCIATICA (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
RESTLESS LEGS SYNDROME (Nervous system disorders) | 3 (3) | 0 (0) | 0 (0)
PARAESTHESIA (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
NEURITIS (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
MIGRAINE (Nervous system disorders) | 1 (1) | 0 (0) | 1 (2)
HYPOAESTHESIA (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
HEADACHE (Nervous system disorders) | 2 (2) | 1 (6) | 0 (0)
DYSKINESIA (Nervous system disorders) | 1 (5) | 0 (0) | 0 (0)
DIZZINESS (Nervous system disorders) | 4 (4) | 0 (0) | 0 (0)
CARPAL TUNNEL SYNDROME (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
BURNING SENSATION (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
INSOMNIA (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
DEPRESSION (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0)
RENAL PAIN (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
POLLAKIURIA (Renal and urinary disorders) | 2 (5) | 0 (0) | 0 (0)
NEPHROLITHIASIS (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
HYPERCALCIURIA (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
HAEMATURIA (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
DYSURIA (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
DYSMENORRHOEA (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
TONSILLAR HYPERTROPHY (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
SINUS CONGESTION (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
RESPIRATORY TRACT CONGESTION (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
COUGH (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (2) | 0 (0)
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
ALLERGIC RESPIRATORY SYMPTOM (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
SKIN REACTION (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 0 (0)
RASH (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
DERMATITIS CONTACT (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0)
DERMATITIS ALLERGIC (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
VARICOSE VEIN (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
HOT FLUSH (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Due to the lack of enrollment, the bone substudy was terminated early.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days